CLINICAL TRIAL: NCT00821886
Title: Phase II Study of Neoadjuvant Ixabepilone/Carboplatin/Trastuzumab in HER2-Positive Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Ixabepilone/Carboplatin/Trastuzumab in HER2-Positive Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 139
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant; Ixabepilone; Carboplatin; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Neoadjuvant Therapy; Trastuzumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone/Trastuzumab/Carboplatin (Experimental): Neoadjuvant treatment with Ixabepilone, Trastuzumab and Carboplatin, followed by surgery, peri-operative treatment and post-operative (adjuvant) treatment if patient deemed to be a surgical candidate
  Interventions: Drug: Ixabepilone; Drug: Trastuzumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Ixabepilone — Ixabepilone 40mg/m2 IV infusion over 3 hours on day 1 of cycles 1-6 (all treatment cycles are 21 days in length)
  Other Names: Ixempra; BMS-247550; NCS 710248; Neoadjuvant Treatment
Drug: Trastuzumab — Trastuzumab 8mg/kg IV over 90 minutes for the first infusion (Cycle 1, Day 1) with a 60 minute post-infusion observation period. Subsequent infusions (Day 1 of Cycles 2-6 with all cycles being 21 days in length) 6mg/kg over 30 minutes if the previous dose was well tolerated; peri-operative trastuzumab 6mg/kg IV every 3-4 weeks; post-operative trastuzumab 6mg/kg IV day 1 every 3 weeks until week 52
  Other Names: Herceptin; Neoadjuvant Therapy
Drug: Carboplatin — Carboplatin AUC=6 IV per institutional guidelines on Day 1 of Cycles 1-6 (all treatment cycles are 21 days in length)
  Other Names: Paraplatin; Neoadjuvant Therapy

SUMMARY:
In this phase II trial the investigators propose to evaluate ixabepilone in combination with carboplatin and trastuzumab as neoadjuvant therapy in locally advanced breast cancer patients. Patients with early stage, HER2-positive breast cancer will receive six cycles of neoadjuvant treatment with ixabepilone, carboplatin, and trastuzumab every three weeks prior to surgery; after surgery, patients will continue treatment with trastuzumab every three weeks until week 52. Concomitant with the post-operative trastuzumab treatment, patients with hormone receptor-positive tumors will receive anti-estrogen treatment. Also, after the completion of chemotherapy, patients may receive radiation treatment at the discretion of their physician.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥18 years of age.
2. Histologically confirmed adenocarcinoma of the breast.
3. Primary palpable disease confined to a breast and axilla on physical examination. For patients without clinically suspicious axillary adenopathy, the primary tumor must be larger than 2 cm in diameter (clinical T2-T3, N0-N1, M0). For patients with clinically suspicious axillary adenopathy, the primary breast tumor can be any size (clinical T1-T3, N1-N2, M0). (T1N0M0 lesions are excluded.)
4. Patients who have no clearly defined palpable breast mass or axillary lymph nodes but are radiographically measurable are eligible. Accepted procedures for measuring breast disease are mammography, MRI, and breast ultrasound. In these patients, radiographic tumor measurements need to be repeated after 3 cycles and prior to surgery.
5. Positive HER2 status (overexpression and/or amplification of HER2 in the primary tumor) as defined by: IHC 3+ or fluorescence in situ hybridization (FISH) positive (ratio >2.2) testing. Documentation of the HER2 results must be available at the time of study enrollment.
6. An ECOG (Eastern Cooperative Oncology Group) performance score of ≤2
7. Normal bone marrow function as defined by:

   * absolute neutrophil count (ANC) >1,500/µL;
   * platelets >100,000/µL;
   * hemoglobin >10 g/dL.
8. Normal hepatic and renal function.
9. Left ventricular ejection fraction (LVEF) within the institutional limits of normal, whichever is lower, as measured by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO).
10. Life expectancy > 12 weeks.
11. Estrogen and progesterone (or estrogen alone) receptor status in the primary tumor known or pending at the time of study enrollment.
12. For women of childbearing potential, negative serum pregnancy test within 7 days prior to starting treatment.
13. For women of childbearing potential, agreement to use a method of contraception that is acceptable to their physician from time of first signing the informed consent until at least 3 months after the last dose of study drug. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately. Patient agreement to discontinue breast-feeding, if applicable, during study treatment. Men enrolled in the study must also agree to use a method of contraception that is acceptable to their physician during their study participation.
14. For patients with previous invasive cancers (including breast cancer) treated with curative intent, completion of chemotherapy or radiation therapy more than 5 years prior to enrollment for this study and no evidence of recurrent disease. Patients may be receiving anti-estrogen hormonal therapy prescribed for previous invasive breast cancer as long as the diagnosis of invasive cancer was made more than 5 years prior to study enrollment. Patients may be using anti-estrogen hormonal therapy at the time of current diagnosis but must discontinue this therapy before beginning study treatment.
15. For patients who had, or will have sentinel lymph node and/or axillary dissection prior to initiation of study treatment, completion at least 4 weeks prior to starting study treatment and well-healed wound.
16. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Previous treatment for this breast cancer.
2. Evidence of metastatic disease.
3. Prior radiation that included ≥30% of major bone marrow-containing areas.
4. Women who are pregnant or breastfeeding.
5. Neuropathy (motor or sensory) ≥grade 1 at study entry.
6. History of significant cardiac disease or cardiac risk factors or the following:

   * uncontrolled arrhythmias
   * poorly controlled hypertension (e.g., systolic blood pressure [BP]> 150 mmHg or diastolic BP >100 mmHg) in spite of optimal medical management
   * angina pectoris requiring antianginal medication or unstable angina within the previous 6 months
   * history of documented congestive heart failure (CHF)
   * any documented myocardial infarction within the previous 6 months
   * clinically significant valvular heart disease
   * current use of medications (e.g., digitalis, beta-blockers, calcium channel-blockers) that alter cardiac conduction, if these medications are administered for the management of cardiac arrhythmia, angina, or CHF. If these medications are administered for other reasons (e.g., hypertension), the patient may be eligible.
   * patients with cardiomegaly on chest x-ray or ventricular hypertrophy on ECG unless ECHO or MUGA scan within the last 3 months demonstrates that the LVEF is ≥ institutional lower limit of normal.
7. Symptomatic intrinsic lung disease.
8. Active malignancy, other than superficial basal cell carcinoma, superficial squamous (skin) cell carcinoma, carcinoma in situ, or non-invasive breast cancer, within the past 5 years.
9. Uncontrolled intercurrent illness including (but not limited to) ongoing or active infection >grade 2.
10. Mental condition or psychiatric disorder rendering the subject unable to understand the nature, scope, and possible consequences of the study or that would limit compliance with study requirements.
11. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving a reasonable suspicion of a disease or condition that contraindicates the use of a study agent or that may affect the interpretation of the results or renders the subjects at high risk from treatment complications.
12. Chronic use of CYP3A4 inhibitors and use of the following strong CYP3A4 inhibitors: ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, amprenavir, indinavir, nelfinavir, delavirdine, and voriconazole. Use of these agents must be discontinued at least 72 hours prior to initiation of study treatment.
13. Received chemotherapy for any indication within the 5 years preceding study enrollment.
14. Prior treatment with trastuzumab or any other anti-HER2 agent for any indication.
15. Concurrent treatment with any other anti-cancer therapy.
16. Concurrent radiation therapy during neoadjuvant study treatment.
17. Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment must be stopped prior to study enrollment.
18. Current therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention of breast cancer. These agents must be discontinued prior to study enrollment.
19. Participation within the previous 30 days in a study with an experimental drug.
20. Known or suspected allergy to Cremophor EL (polyoxyethylated castor oil), a drug formulated in Cremophor EL such as paclitaxel, or any other agent given in the course of this trial.
21. Inability or unwillingness to comply with study procedures including those for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Started | 58 (Two patients were enrolled, but subsequently found to be ineligible)
Completed | 49
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 53 [25 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: Proportion of patients who do not exhibit residual invasive breast cancer in breast or axillary lymph nodes at time of surgery
Time Frame: average18 months
Population: Patients who underwent surgery per protocol
Measure: Number; unit: participants
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Number analyzed (Participants) | 52
participants | 27

2. Secondary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Toxicity
Description: Assessment based on the frequency of treatment-related adverse events according to NCI CTCAE criteria v3.0.
Time Frame: Day 1 of each 3 week cycle up to 6 cycles , and every 9 weeks post-surgery until treatment discontinuation
Population: Includes eligible patients
Measure: Number; unit: participants
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Number analyzed (Participants) | 58
participants
  Fatigue | 54
  Anemia | 50
  Neutropenia | 49
  Peripheral neuropathy | 47
  Leukopenia | 46
  Nausea | 45
  Thrombocytopenia | 40
  Alopecia | 26
  Diarrhea | 25
  Constipation | 21
  Anorexia | 19
  Vomiting | 18
  Arthralgia | 16
  Dyspnea | 14
  Myalgia | 14
  Pain - extremity | 14
  Dysgeusia | 13
  GERD | 13
  Rash | 13
  Edema | 12
  Febrile neutropenia | 4

3. Secondary Outcome: Disease-free Survival
Description: Defined as the interval from the first date of study treatment until the date of tumor recurrence or death from any cause
Time Frame: expected average 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Number analyzed (Participants) | 58
months | NA [53.03 to NA] — Median DFS and upper 95% CI not reached at this time point

4. Secondary Outcome: Overall Survival
Description: Defined as the time between Day 1 Cycle 1 to date of death from any cause.
Time Frame: approximately 48 months
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Number analyzed (Participants) | 58
months | NA [NA to NA] — Median OS and 95% CI not reached at this time point

ADVERSE EVENTS:
Description: Adverse Event analysis includes patients who were enrolled and treated
Arm/Group | Ixabepilone/Trastuzumab/Carboplatin
Serious Adverse Events (participants affected / at risk) | 17/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone/Trastuzumab/Carboplatin (N=58)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4
Infections and infestations - Other, MRSA (Infections and infestations) | 2
Bronchial infection (Infections and infestations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Fetal Death (Pregnancy, puerperium and perinatal conditions) | 1
Fever (General disorders) | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1
Infections and infestations - Other, surgical incision site infection (Infections and infestations) | 1
Non-cardiac chest pain (General disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Skin infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone/Trastuzumab/Carboplatin (N=58)
Fatigue (General disorders) | 54
Anemia (Blood and lymphatic system disorders) | 50
Neutrophil count decreased (Blood and lymphatic system disorders) | 49
Peripheral sensory neuropathy (Nervous system disorders) | 47
White blood cell decreased (Blood and lymphatic system disorders) | 46
Nausea (Gastrointestinal disorders) | 45
Platelet count decreased (Blood and lymphatic system disorders) | 40
Alopecia (Skin and subcutaneous tissue disorders) | 26
Diarrhea (Gastrointestinal disorders) | 25
Constipation (Gastrointestinal disorders) | 21
Anorexia (Metabolism and nutrition disorders) | 19
Vomiting (Gastrointestinal disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Dysgeusia (Nervous system disorders) | 13
Gastroesophageal reflux disease (Gastrointestinal disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 13
Edema (General disorders) | 12
Hot flashes (Vascular disorders) | 11
Headache (Nervous system disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Insomnia (Psychiatric disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 8
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7
Mucositis (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 7
Paresthesia (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Upper respiratory infection (Infections and infestations) | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Chills (General disorders) | 5
Fever (General disorders) | 5
Pain (General disorders) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blurred vision (Eye disorders) | 4
Depression (Psychiatric disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Non-cardiac chest pain (General disorders) | 4
Oral pain (Gastrointestinal disorders) | 4
Alkaline phosphatase elevated (Investigations) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 3
Infection at port site (Infections and infestations) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, throat pain (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Eye disorders - Other, vision changes (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites